CLINICAL TRIAL: NCT04891848
Title: Assessment of Inflammation With Haematological Parameters in Patients With Migraine and Tension Type Headache: a Prospective Study From a Tertiary Care Center
Brief Title: Assessment of Inflammation in Primary Headaches
Status: Completed | Type: Observational
Sponsor: Kocaeli University (Other)
Responsible Party: Principal Investigator, Halil Okay Albayrak, Principal Investigator, Department of Emergency Medicine, Kocaeli University
Other Study IDs: KOU/KAE: 2018/192
Record Dates: First submitted 2021-04-20; First posted 2021-05-19 (Actual); Last update posted 2021-05-19 (Actual); Status verified 2021-05

CONDITIONS: Headache Disorders
Keywords: primary headache; migraine with aura; migraine without aura; tension type headache; inflammation; neuroinflammation
MeSH Terms: conditions — Headache Disorders; Migraine with Aura; Migraine without Aura; Tension-Type Headache; Inflammation; Neuroinflammatory Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- migraine with aura: 51 patients with MA
  Interventions: Other: inflammation
- migraine without aura: 51 patients with migraine without aura
  Interventions: Other: inflammation
- tension type headache: 48 patients with tension type headache
  Interventions: Other: inflammation
- healthy controls: 80 healthy participants
  Interventions: Other: inflammation

INTERVENTIONS:
Other: inflammation — inflammatory values in complete blood count (CBC)

SUMMARY:
Headache is the most common neurological complaint accounting for % 1 to % 4 in the emergency department (ED).Every year, nearly one million people with headache attacks have been consulted by healthcare professionals at the emergency room in the United States.The International Classification of Headache Disorders (ICHD) divided headaches into two main groups: primary headaches and secondary headaches. The vast majority of cases who presented with acute headache attack in ED had a diagnosis of primary headache disorders (tension- type headache, migraine, cluster- type headache, and other primary headaches). However, secondary headache is often associated with underlying intracranial pathologies, and noted in % 10 of cases in emergency rooms. Despite the frequent presence of primary headaches, limited time setting and busy periods of medical assessment, leading diagnostic and therapeutic options due to the pathophysiological factors to be overlooked.

To date, no study in the emergency care setting has explored the role of inflammation in patients with acute migraine and TTH. Investigators aimed to explore inflammatory markers [white blood cells (WBC), neutrophil, lymphocyte, platelet, neutrophil / lymphocyte ratio (NLR), and platelet / lymphocyte ratio (PLR)] in complete blood count (CBC) among MA, MO, and TTH participants who admitted to ED with acute headache attack and healthy volunteers.

DETAILED DESCRIPTION:
Study design This prospective study was completed at an emergency care of a tertiary referral hospital between May 2018 and May 2019. The hospital admits a total of 45.000 adult emergency patients per year. This study was approved by the local ethics Committee of Kocaeli University (KOU/KAE: 2018/192) in accordance with the Helsinki Declaration. Written and informed consent form was obtained from all individual participants.

Study population Investigators screened 720 patients who admitted to the ED with an acute headache attack. Clinical evaluation was performed by an experienced neurologist. Consequently, 51 patients with MA, 51 patients with MO, and 48 patients with TTH according to the diagnostic criterias of ICHD-3 and 80 age- and gender matched healthy controls were enrolled in this study. Detailed sociodemographic and clinical data collected using face-to-face interview. Visual analog scale (VAS) documented to measure the intensity of pain in patient groups.

Investigators included adult participants aged between 18 and 65 years. Also, subjects were eligible for inclusion if their body mass index (BMI) ranges were between18 kg/m2 and 30 kg/m2. Patients with secondary headaches, trauma, malignancy, chronic inflammatory disorders, infectious diseases, hematologic abnormalities, a prior history of surgery (within the preceding 6 months), receiving analgesics, antibiotics, blood transfusion and other blood products, were excluded from the study.

Laboratory analysis Complete blood count (CBC) parameters [WBC, neutrophil, lymphocyte, platelet] of patients and control groups were obtained from 2 cc peripheral venous blood samples (purple K3 EDTA tubes, Beckman Coulter DXH 800 Analyzer) during admission. NLR and PLR were calculated by dividing absolute neutrophil to absolute lymphocyte count and absolute platelet to absolute lymphocyte count, respectively.

Statistical Analysis SPSS 17.0 statistical software package program (IBM Corporation, USA) was used for the analysis. Descriptive data were presented using numbers, percentages (%) , mean ± standard deviation. Categorical variables were analyzed by using chi-square (χ2) test. Normality tests (Shapiro-Wilks, Lilliefors, and Kolmogorov-Smirnov) were used for all parameters. Due to the non-normal distribution of CBC values, Kruskal-Wallis and Tamhane's T2 post hoc tests were used to compare between patients with MA, MO, TTH, and healthy controls. A p value ≤ 0.05 considered statistically significant.

ELIGIBILITY:
Inclusion Criteria;

* Clinical diagnosis of Migraine
* Clinical diagnosis of Tension- type headache
* Age between 18 and 65 years
* Body mass index between 18 kg/m2 and 30 kg/m2

Exclusion Criteria;

* Secondary headaches
* Chronic inflammatory disorders
* Infectious diseases
* Hematologic abnormalities
* A prior history of surgery (within the preceding 6 months)
* Receiving analgesics
* Blood transfusion before admission

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Migraine and tension-type headache patients who admitted to emergency department with an acute headache attack
Sampling Method: Non-Probability Sample
Enrollment: 230 (Actual)
Dates: Start 2018-05-01 (Actual); Primary Completion 2019-05-31 (Actual); Study Completion 2019-05-31 (Actual)

PRIMARY OUTCOMES:
White blood cells | Up to 1 year
  White blood cells (x10³/μL) counted in complete blood count and compared between patients and healthy controls
Neutrophil | Up to 1 year
  Neutrophil (x10³/μL) levels counted in complete blood count and compared between patients and healthy controls
Lymphocyte | Up to 1 year
  Lymphocyte (x10³/μL) levels counted in complete blood count and compared between patients and healthy controls
Platelet | Up to 1 year
  Platelet (x10³/μL) levels counted in complete blood count and compared between patients and healthy controls
Neutrophil/lymphocyte ratio | Up to 1 year
  Neutrophil/lymphocyte ratio calculated by dividing absolute neutrophil to absolute lymphocyte and compared between patients and healthy controls.
Platelet/lymphocyte ratio | Up to 1 year
  Platelet/lymphocyte ratio calculated by dividing absolute platelet to absolute lymphocyte and compared between patients and healthy controls.

CONTACTS AND LOCATIONS:
Overall Officials: Serkan Yılmaz, Prof, Study Chair — Kocaeli University Department of Emergency Medicine; Serkan Yılmaz, Prof, Study Director — Kocaeli University Department of Emergency Medicine
Locations (1):
- Halil Okay Albayrak, Kocaeli, İzmit, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Albayrak HO, Gurbuz H, Basaran S, Yilmaz S. Assessment of inflammation with hematological parameters in patients with migraine and tension-type headache: a prospective study from a tertiary care center. Pain Manag. 2022 Mar;12(2):141-148. doi: 10.2217/pmt-2021-0036. Epub 2021 Aug 25. PMID 34431322